CLINICAL TRIAL: NCT07193589
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study Evaluating the Efficacy and Safety of ZL-82 Tablets in Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase II Clinical Study Evaluating of ZL-82 Tablets in Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL-82-AD-II
Record Dates: First submitted 2025-04-27; First posted 2025-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: ZL-82
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The high-dose group of ZL-82 tablets (Experimental)
  Interventions: Drug: The high-dose group of ZL-82 tablets
- The low-dose group of ZL-82 tablets (Experimental)
  Interventions: Drug: The low-dose group of ZL-82 tablets
- The placebo group (Placebo Comparator)
  Interventions: Drug: The placebo group

INTERVENTIONS:
Drug: The high-dose group of ZL-82 tablets — Participants will take the investigational drug orally for 16 weeks, 200mg each time , once a day.
  Arms: The high-dose group of ZL-82 tablets
Drug: The low-dose group of ZL-82 tablets — Participants will take the investigational drug orally for 16 weeks, 100mg each time, once a day.
  Arms: The low-dose group of ZL-82 tablets
Drug: The placebo group — The participants will take the investigational drug orally for 16 weeks, 2 tablets each time , once a day.
  Arms: The placebo group

SUMMARY:
This clinical trial aims to explore whether the drug ZL-82 tablets can be used to treat moderate to severe atopic dermatitis in adults, and to understand the safety and tolerability of the drug. The main questions that the trial intends to answer are: Can ZL-82 tablets alleviate the Eczema Area and Severity Index (EASI) score of patients? What physical problems will patients have after taking ZL-82 tablets? The researchers will compare ZL-82 tablets with placebo (a substance with a similar appearance but without drug components) to observe whether ZL-82 tablets can be used to treat moderate to severe atopic dermatitis. Participants need to take ZL-82 tablets or placebo every day for 16 weeks, and visit the hospital for a check-up every two weeks; record their own symptoms and the percentage change of EASI score relative to the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged 18 years and above and 75 years and below (inclusive of the threshold value, based on the date of signing the ICF), with BMI >= 19 kg/m2.
2. Participants are fully informed of the purpose and requirements of this trial, and voluntarily sign the informed consent form.
3. According to the Hanifin & Rajka diagnostic criteria (≥ 3 out of 4 main 4, >= 3 out of 23 secondary symptoms, see Appendix 1), diagnosed as AD by the investigators, and with a history of AD for >= 1 year before screening.

4 . The definition of moderate to severe atopic dermatitis during screening and baseline period is as follows:

1. IGA score of 3 or 4;
2. EASI score >= 16;
3. Average peak pruritus NRS score >= 4 in the past week (Note: The NRS average value is the average of the maximum NRS score of pruritus intensity over 7 consecutive days before baseline, with a score range of 0-10 for each day. At least 4 days of scores are required for the calculation of the average score);
4. BSA (body surface area) affected by AD >= 10% (BSA: body surface area, in this trial, BSA is based on the average human body surface area of 1.6 m2); 5. Participants who have been treated with local corticosteroid drugs, calcineurin inhibitors, or phototherapy within the past 6 months, and whose medical history indicates inadequate response, no response, or intolerance to these treatments, or who have medical contraindications for such treatments (treatment duration ≥ 4 weeks), and who require systemic treatment to control the disease, should be selected. Note: For stable treatment response that is insufficient when using local drugs (such as moderate-to-high potency topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI)), insufficient response is defined as participants receiving treatment for the recommended duration or the maximum recommended duration as per the instructions, but failing to achieve and maintain disease remission (corresponding to IGA score = 0 [clear] - 2 [mild]).

   6. Use a mild moisturizing agent (moisturizing cream) at a stable dose twice a day for at least 7 consecutive days before the first day of administration, and agree to continue using it during the study.

Exclusion Criteria:

1. Allergy to the test drug or any component thereof, or allergy or intolerance to other oral Janus kinase (JAK) inhibitors.
2. Use of any of the following drugs or treatments:

   a. Within 1 month before the baseline, received other oral JAK inhibitor treatment, or had a lack of efficacy or intolerance to other oral JAK inhibitors, including but not limited to baricitinib, upadacitinib, abrocitinib, etc.; b. Within 6 weeks before the baseline, used upadilunab/spicibaydin; c. Within 3 months before the baseline (or within 5 drug half-lives, whichever is longer), used other systemic biological agents known or potentially affecting AD other than dupilumab (such as IL-13 receptor antibody [crizorilumab], IL-31Rα antibody [nimotuzumab] etc.); d. Within 1 week before the baseline, used any AD topical treatment: TCS, TCI, PDE-4 inhibitor, JAK inhibitor, traditional Chinese medicine / Chinese patent medicine, herbal medicine, etc.; e. Within 4 weeks before the baseline (or within 5 half-lives, whichever is longer), used any systemic treatment for AD: immunosuppressants (such as cyclosporine, methotrexate, azathioprine, mycophenolate mofetil, etc.), glucocorticoids, PDE-4 inhibitor, etc.; f. Within 4 weeks before the baseline received any systemic treatment for AD or other autoimmune inflammatory diseases, common AD herbal medicine preparations or Chinese patent medicines; g. Within 4 weeks before the baseline received phototherapy (narrow-band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), sunbed or any other light-emitting device treatment; h. Within 6 months before the baseline received allergen-specific immunotherapy; i. Within 2 weeks before the baseline or within 5 half-lives of the drug (whichever is longer), systemically used (or expected to be needed throughout the study period) strong or moderate inhibitors or inducers of cytochrome P450 (CYP) (see Appendix II); j. Within 2 weeks before the baseline or within 5 half-lives of the drug (whichever is longer), systemically used (or expected to be needed throughout the study period) P-glycoprotein (P-gp) inhibitors (see Appendix II); k. Had received lymphocyte depletion therapy before (such as: alegrucilunab, anti-CD4 drugs, cladribine, rituximab, omalizumab, cyclophosphamide, mitoxantrone, total body irradiation, bone marrow transplantation, darzalex); l. Within 3 months before the baseline or within 5 half-lives of the drug (if known, whichever is longer), received any treatment in clinical studies of drugs or medical devices, or was currently enrolled in another interventional study.
3. Individuals with a history of major diseases: This includes but is not limited to those with a history of diseases in the digestive system, cardiovascular system, respiratory system, musculoskeletal system, endocrine system, nervous and mental system, hematological system, immune system disorders, thromboembolic diseases (or individuals at high risk of thromboembolism), and metabolic abnormalities, or those who have undergone major surgeries, or any other diseases or physiological conditions that the investigator deems may affect the trial results.
4. Family Planning: a. Pregnant or lactating women; b. Throughout the entire study period, all participants or their spouses (or partners) who have reproductive capacity must ensure to take effective contraceptive measures from the moment of signing the informed consent form until 90 days after the last administration of the drug (contraceptive measures and requirements are detailed in Appendix III); c. Those who plan to donate eggs or sperm during the trial period and within 3 months after the last administration.
5. Those who have a history of malignant tumors in the past, including solid tumors and hematological malignancies (excluding basal cell carcinoma and cutaneous squamous cell carcinoma that have been removed or cured).
6. Those who have undergone major surgical procedures within 4 weeks before screening or are scheduled to undergo such procedures during the screening period.
7. Those whose hepatitis B surface antigen or hepatitis B core antibody (except for HBV DNA results within the normal range) is positive, hepatitis C antibody (except for HCV RNA results within the normal range) is positive, human immunodeficiency virus antibody is positive, or Treponema pallidum antibody is positive (excluding those with negative RPR/TRUST test results).
8. Participants should have resting systolic blood pressure (SBP) < 90 mmHg and/or diastolic blood pressure (DBP) < 55 mmHg before the first administration. Participants with hypertension (SBP >= 160 mmHg, DBP >= 100 mmHg) treated with two or more antihypertensive drugs but with poor control, and those with severe sleep apnea and other diseases, and those judged by the investigators to have conditions that may interfere with the clinical trial results or affect the safety of the participants.
9. 12-lead ECG before screening and before the first administration suggests that the PR interval > 200 msec, heart rate < 55 bpm, and corrected Fridericia QT interval (QTcF) >= 450 ms (for males), and >= 470 ms for females. 10. Participants with a history of severe cardiovascular and cerebrovascular diseases and poor control, including myocardial infarction, unstable angina pectoris, congestive heart failure, congenital heart disease, stroke or transient ischemic attack; and those with bleeding tendencies, or who have had intracerebral hemorrhage within the past 1 year.

11. Those with any of the following medical histories:

a. Symptoms of bradycardia or related medical history; b. Second or third degree atrioventricular block; c. Cardiac arrest duration > 3 seconds; d. History of sick sinus syndrome or neurocardiac syncope. 12. Those with a history of uncontrolled diabetes (defined as HbA1c > 9%). 13. Those with any systemic disease that may affect the evaluation of the trial results or active other skin diseases (such as psoriasis, lupus erythematosus, Netherton syndrome, chronic actinic dermatitis, dermatitis herpetiformis), or those with scars, freckles, tattoos, obvious pigmentation and other factors that may affect the evaluation of skin lesions at the affected sites.

14. Those with >= 2 grade peripheral neuropathy according to CTCAE V5.0 during screening, and those with any significant neurological dysfunction remaining.

15. Those with a history of current active primary or secondary immunodeficiency diseases.

16. Those with previous disseminated herpes zoster or herpes simplex. 17. Those with a history of significant pulmonary diseases such as chronic obstructive pulmonary disease, pulmonary fibrosis, severe or poorly controlled asthma (except for mild intermittent asthma that does not require routine maintenance treatment).

18. Select patients who need intravenous antibiotics for hospitalization within the past 30 days or who need oral antibiotic treatment for active bacterial, fungal, viral, mycobacterial infections or other infections within the past 14 days before screening.

19. Select patients who have received any live or attenuated vaccines within the past 30 days before screening or who plan to receive any live or attenuated vaccines during the study period or within 30 days after the last administration.

20. Select patients who have a history of active tuberculosis within the past 1 year before screening or who have a positive tuberculosis test result within the past 1 month before screening. These are defined as:

a. Have a history of active tuberculosis infection and no evidence of clinical cure; b. Have imaging evidence (such as chest CT) indicating active tuberculosis in the subject at the time of screening; c. Have suspicious tuberculosis symptoms that cannot be excluded by the investigator's assessment (such as low fever, cough, night sweats, weight loss, etc.); d. Latent tuberculosis infection (LTBI): Have a positive tuberculosis test result during the screening period, but no clinical symptoms or signs of active tuberculosis; Detection methods include but are not limited to T-spot test, QuantiFERON-TB Gold test, PPD test. If the subject has started LTBI preventive treatment according to the guideline-approved protocol before randomization and has been treated for at least 1 month, the subject is eligible. To continue the study, the subject must agree to complete the recommended treatment course for LTBI; e. The result of the tuberculosis test: If the result of the first test is uncertain, a second test should be conducted. If the retest result is still uncertain, the subject should be excluded from this study. If the retest is positive, the subject should receive LTBI treatment. If the retest is negative and does not meet other tuberculosis exclusion criteria, the subject is eligible.

21. During the screening visit, abnormal results of blood routine tests were screened (repeated tests could be conducted for verification, and the decision was made independently by the researchers). The abnormalities included, but were not limited to:

a. White blood cell count < 3.5 × 10^9/L; b. Neutrophil count < 1.5 × 10^9/L; c. Lymphocyte count < 0.8 × 10^9/L; d. Platelet count < 100 × 10^9/L; e. Hemoglobin < 9.0 g/dL. 22. During the screening visit, abnormal results of blood biochemistry (repeated tests are allowed for verification, and the determination is made independently by the researchers), including but not limited to:

1. Total bilirubin > 1.5 × upper limit of normal (ULN);
2. AST > 1.5 × ULN;
3. ALT > 1.5 × ULN. 23. With moderate or end-stage renal function impairment, including but not limited to:

a. Estimated glomerular filtration rate < 60 mL/min/1.73 m2; b. Estimated creatinine clearance rate < 60 mL/min; c. Creatinine level > 1.4 mg/dL or 123 μmol/L (for female participants); d. Creatinine level > 1.6 mg/dL or 141 μmol/L (for male participants). 24. Exclude participants who have a history of alcohol abuse within the past 1 year (with weekly alcohol intake exceeding 21 units for men and 14 units per week for women (1 unit = 360 mL of beer; or 150 mL of wine; or 45 mL of liquor)) or a history of drug abuse.

25. Accept those who have received any of the following treatments:

1. Within 12 weeks before the first administration of the investigational drug:

   1. Intravenous immunoglobulin or plasma exchange therapy;
   2. Drugs known to have an impact on the cardiac conduction system (such as Class I or III anti-arrhythmic drugs);
   3. Other biologics except dupilumab.
2. Within 4 weeks before administration, those who have used long-acting anticoagulant drugs (such as warfarin, dabigatran, etc.) or those who need continuous anticoagulant drug treatment (except aspirin <= 100 mg/day).
3. Within 1 week before the first administration of the investigational drug.

   1) Use antiplatelet drugs. Note: Based on the investigator's judgment, low-dose aspirin (dose <= 100 mg, QD) for the purpose of preventing cardiovascular diseases is allowed; 26. Within 12 weeks before screening, those who have lost blood >= 400 mL (including trauma, blood collection, blood donation), or those who plan to donate blood during the study or within 1 month after the study.

   27. Due to other reasons, unable to complete this study or considered unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the percentage changes in Eczema Area And Severity Index (EASI) scores from baseline between the ZL-82 tablets dose group and the placebo group. | At the 16th week

SECONDARY OUTCOMES:
Compare respectively the percentage changes of EASI scores from baseline in the ZL-82 tablets dose group and the placebo group | At the 2nd, 4th, 8th and 12th weeks
Compare respectively the proportions of participants in the ZL-82 tablets dose group and the placebo group whose EASI scores have improved by at least 50% (EASI-50), 75% (EASI-75) and 90% (EASI-90). | At the 2nd, 4th, 8th and 12th weeks
Compare respectively the proportions of participants in the ZL-82 tablets dose group and the placebo group who had an IGA score of 0 or 1 and showed a 2-point improvement compared to the baseline in the Investigator's Global Assessment (IGA) method. | At the 2nd, 4th, 8th, 12th and 16th weeks
Compare the proportions of participants whose IGA scores improved by ≥ 2 points relative to the baseline in the ZL-82 tablet dose group and the placebo group respectively. | At the 2nd, 4th, 8th, 12th and 16th weeks
The weekly average peak pruritus numerical rating scale (PPNRS) scores of the ZL-82 tablets dose group and the placebo group were compared respectively to evaluate the changes from baseline. | At the 2nd, 4th, 8th, 12th and 16th weeks
Compare respectively the proportions of participants whose weekly average PPNRS scores relative to the baseline were ≥ 4 points in the ZL-82 tablets dose group and the placebo group. | At the 2nd, 4th, 8th, 12th and 16th weeks
Compare respectively the changes in the body surface area (BSA) affected by AD relative to the baseline in the ZL-82 tablets dose group and the placebo group. | At the 2nd, 4th, 8th, 12th and 16th weeks
The changes in Dermatology Life Quality Index (DLQI) relative to the baseline were compared respectively between the ZL-82 tablets dose group and the placebo group. | At the 2nd, 4th, 8th, 12th and 16th weeks
The changes in the scores of the Patient-Oriented Eczema Measure (POEM) scale, a self-assessment scale for eczema, of the participants in the ZL-82 tablets dose group and the placebo group relative to the baseline were compared respectively. | At the 2nd, 4th, 8th, 12th and 16th weeks
health checkup | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141.If necessary, planned external visits to the participants must be conducted.
vital signs | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141.If necessary, planned external visits to the participants must be conducted.
  body temperature
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  White blood cell
laboratory tests results | Screening period,Day141.If necessary, planned external visits to the participants must be conducted.
  urobilinogen
PR interval | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
ZL-82 tablets blood drug concentration-time curve | Day1 Within 30 minutes before administration and 5minutes，15 minutes ，0.5 hours，1 hours，1.5 hours，2 hours，3 hours，4 hours，6 hours，8 hours after administration, Day15,Day29,Day57,Day85,Day113.
PK parameters of ZL-82 tablets in blood(Cmax ) | Day1 Within 30 minutes before administration and 5minutes，15 minutes ，0.5 hours，1 hours，1.5 hours，2 hours，3 hours，4 hours，6 hours，8 hours after administration
The steady-state plasma concentration (Cmin, ss) of ZL-82 tablets before administration (Pre-dose) | Day1,Day15,Day29,Day57,Day85,Day113,If necessary, planned external visits to the participants must be conducted.
vital signs | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141.If necessary, planned external visits to the participants must be conducted.
  blood pressure
vital signs | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141.If necessary, planned external visits to the participants must be conducted.
  respiration
vital signs | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141.If necessary, planned external visits to the participants must be conducted.
  pulse
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Red blood cell
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  platelet count
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Neutrophil granulocyte
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Total Protein
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Albumin
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  total bilirubin
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  direct bilirubin
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  indirect bilirubin
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  globulin
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  alkaline phosphatase
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  total cholesterol
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  triglycerides
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  high-density lipoprotein
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Low Density Lipoprotein
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  fasting blood-glucose
laboratory tests results | Day-28 to Day-1,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  creatinine
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  urea nitrogen
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  Uric Acid
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  coagulation function
laboratory tests results | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
  urine test
QRS interval | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
QT/QTc interval | Screening period,Day1,Day15,Day29,Day57,Day85,Day113,Day141,If necessary, planned external visits to the participants must be conducted.
PK parameters of ZL-82 tablets in blood(Tmax) | Day1 Within 30 minutes before administration and 5minutes，15 minutes ，0.5 hours，1 hours，1.5 hours，2 hours，3 hours，4 hours，6 hours，8 hours after administration
adverse event | From date of randomization until the date of completion of data collection, assessed up to 20 weeks
  Adverse events, serious adverse events, suspected and unexpected serious adverse reactions (SUSAR), priority adverse reactions, incidence of adverse reactions

OTHER OUTCOMES:
Eosinophil count | Day1,Day15,Day29,Day57,Day85,Day113,If necessary, planned external visits to the participants must be conducted.
  Evaluate the changes in PD biomarkers of ZL-82 tablets in participants with moderate to severe AD.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No